CLINICAL TRIAL: NCT02164942
Title: LCI-GU-BLA-SPEC-001: Expression of the Aurora Kinase Family and Chemoresistance in Muscle-Invasive Bladder Cancer
Brief Title: LCI-GU-BLA-SPEC-001: Aurora Kinase Expression in Muscle-Invasive Bladder Cancer
Status: Terminated | Type: Observational
Why Stopped: Futility
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Other Study IDs: LCI-GU-BLA-SPEC-001; 00009729
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2017-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single Arm: Specimen Collection

SUMMARY:
This is a prospective, single arm, observational study examining aurora kinases and circulating tumor cells in subjects with bladder cancer being treated with standard cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
Subjects will receive neoadjuvant cisplatin-based chemotherapy followed by radical cystectomy per standard of care. CTC and Aurora kinase expression patterns will be analyzed in subject specimens for correlation with clinicopathologic outcome. Subjects will be on study for a total of five years following cystectomy.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed American Joint Committee on Cancer seventh edition clinical stage T2-4a N0-3 urothelial carcinoma of the bladder based on diagnostic transurethral bladder biopsy or transurethral resection of bladder tumor (TURBT) confirming the presence of urothelial carcinoma with muscularis propria invasion.
* Archived tissue from prior biopsy/resection must be available for baseline AK analysis.
* Subjects must be eligible to undergo radical cystectomy and cisplatin-based chemotherapy.
* Subjects with radiographically enlarged lymph nodes (short axis >10 mm with CT scan or MRI) should undergo percutaneous biopsy for staging in accordance with local practices, though preferred, is not mandatory for study enrollment.
* A baseline computed tomography (CT) scan with intravenous contrast of the chest, abdomen and pelvis is required in all subjects. A radionuclide bone scan is also required in subjects with skeletal pain or abnormally elevated alkaline phosphatase values.
* Age at least 18 years old.
* ECOG performance status of 0 or 1.
* Bilirubin less than 1.5 mg/dL.
* Subjects must have adequate liver function: AST and ALT less than 2.5x upper limit of normal, alkaline phosphatase less than 2.5x upper limit of normal.
* Subjects must have adequate bone marrow function: Platelets greater than 100,000 cells/mm3, Hemoglobin greater than 9.0g/dL and ANC greater than 1,500 cells/mm3.
* Subjects must have adequate renal function with creatinine clearance of at least 60 mL/min.
* Subjects must sign a written informed consent document and authorization for release of their medical records for the purposes of research.

Exclusion Criteria

* Pure non-urothelial or mixed small cell histology identified within TURBT specimen.
* Absence of documented urothelial carcinoma with muscularis propria invasion on diagnostic transurethral bladder biopsy or transurethral resection of bladder tumor (TURBT).
* Distant metastatic disease, including non-regional lymphadenopathy and visceral metastases, identified on pretreatment radiographic studies.
* Creatinine clearance less than 60 mL/min.
* CTCAE version 4 grade 2 or greater hearing loss.
* CTCAE version 4 grade 2 or greater peripheral neuropathy.
* NYHA class III heart failure or cardiac ejection fraction less than or equal to 50%.
* Women of child-bearing age who are pregnant or breast feeding.
* Uncontrolled and current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with other active malignancies as defined as synchronous malignancy at the time of bladder cancer diagnosis, excluding non-metastatic, non-melanoma skin cancer are excluded.
* Major surgery within 4 weeks of consent.
* Subjects requiring therapeutic anticoagulation at the time of consent.
* Currently enrolled on another clinical trial for the treatment of bladder cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with muscle-invasive urothelial carcinoma of the bladder
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Correlation of pathologic response rate and aurora kinase expression | Within 6 months of subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Tesa M Adams, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Healthcare System, Charlotte, North Carolina, United States